CLINICAL TRIAL: NCT00480597
Title: Randomised, Multicenter Phase II Study in Patients With Metastatic Breast Cancer With Gemcitabine Plus Vinorelbine Versus Gemcitabine Plus Cisplatin Versus Gemcitabine Plus Capecitabine
Brief Title: Gemcitabine/Vinorelbine Versus Gemcitabine/Cisplatin Versus Gemcitabine/Capecitabine in Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Gemcitabin 02 MC
Record Dates: First submitted 2007-05-30; First posted 2007-05-31 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2007-05

CONDITIONS: Metastatic Breast Cancer
Keywords: gemcitabine; vinorelbine; cisplatin; capecitabine; pretreated metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Cisplatin; Vinorelbine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: gemcitabine
Drug: cisplatin
Drug: vinorelbine
Drug: capecitabine

SUMMARY:
Development of an active second-line treatment option for metastatic breast cancer patients previously pre-treated with anthracyclines and taxanes in neoadjuvant, adjuvant or palliative settings.

For each randomisation arm, 47 patients will be included. The trial was performed as a 2-stage phase II study according to the optimal design by Simon with overall response rate as the primary objective.

Study Design:

Arm A Gemcitabine 1000 mg/m2 d1, 8; Vinorelbine 25 mg/m2 d1, 8 q 3 weeks

Arm B Gemcitabine 1000 mg/m2 d1, 8; Cisplain 30 mg/m2 d1, 8 q 3 weeks

Arm C Gemcitabine 1000 mg/m2 d1, 8; Capecitabine 1650 mg/m2 oral d1-14 q 3 weeks

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic breast cancer
* All patients were required to give written informed consent
* Only one prior chemotherapy for metastatic breast cancer was allowed. This clinical trial was designed to test the efficacy of a second-line chemotherapy.
* Antracycline-pretreatment during aduvant or palliative first line therapy
* Bidimensionally measurable lesion outside a previous radiation field.
* Age >= 18 years
* Karnofsky Performance status >= 70%
* Adequate heamatological, renal, cardiac and hepatic function
* No radiation of the measurable lesion during the study was allowed.

Exclusion Criteria:

* Only bone metastases
* Active infection
* Previous treatment with one of the study drugs
* Application of other cytotoxic chemotherapy
* Insufficent renal function (creatinine clearance < 60ml/min)
* Known DPD deficiency
* clinically unstable brain metastasis
* pregancy or lactation
* other primary malignancies (other than carcinoma-in-situ of the cervix or adequately treated basal cell cancer of the skin).

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2002-10

PRIMARY OUTCOMES:
Response rate | one year after last patient in

SECONDARY OUTCOMES:
Time to progression | one year after last patient in
Overall Survival | one year after last patient in
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Volker Heinemann, PhD, MD, Principal Investigator — University of Munich - Klinikum Grosshadern

REFERENCES:
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241